CLINICAL TRIAL: NCT00932646
Title: Characterization of 24 Hour Spirometry Profiles of Inhaled BI 1744 CL and Inhaled Foradil in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Characterisation of 24-hour FEV1-time Profiles of Inhaled BI 1744 CL and Inhaled Foradil in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.25
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Formoterol Fumarate

ARMS (4):
- BI1744 (Olodaterol) (Experimental): Medium Dose once Daily
  Interventions: Drug: BI 1744 (Olodaterol) Medium Dose
- BI 1744 (Olodaterol) (Experimental): Low Dose once Daily
  Interventions: Drug: BI 1744 (Olodaterol) Low Dose
- Placebo (Placebo Comparator): Placebo once Daily
  Interventions: Drug: Placebo
- Foradil (Active Comparator): 12 mcg twice daily
  Interventions: Drug: Foradil

INTERVENTIONS:
Drug: BI 1744 (Olodaterol) Low Dose — BI1744 Respimat low dose once daily and placebo Foradil
  Arms: BI 1744 (Olodaterol)
Drug: BI 1744 (Olodaterol) Medium Dose — BI1744 Respimat medium dose once daily and placebo Foradil
  Arms: BI1744 (Olodaterol)
Drug: Placebo — Placebo Respimat once daily and placebo Foradil
  Arms: Placebo
Drug: Foradil — 12 mcg twice daily and placebo Respimat
  Arms: Foradil

SUMMARY:
The study is intended to characterize the lung function profile of BI1744 in COPD patients where patients will perform pulmonary function tests at regular intervals for 24 hours at the end of a 6 week treatment period. Each patient will receive all four treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate with confirmed diagnosis of COPD
* 40 years of age or older
* having a 10 pack year smoking history
* able to perform serial pulmonary function tests
* able to use both a DPI and Respimat device

Exclusion Criteria:

Significant other disease

* clinically relevant abnormal hematology, chemistry, or urinalysis
* history of asthma
* diagnosis of thyrotoxicosis
* paroxysmal tachycardia related to beta agonists
* history of MI within 1 year, cardiac arrhythmia, hospitalization for heart failure within 1 year
* active tuberculosis, cystic fibrosis, clinically evident bronchiectasis
* significant alcohol or drug use
* pulmonary resection
* taking oral beta adrenergics
* taking unstable oral steroids
* daytime oxygen
* enrolled in rehabilitation program
* enrolled in another study or taking investigational products
* pregnant or nursing women, women of child bearing potential not willing to use two methods of birth control
* those who are not willing to comply with pulmonary medication washouts

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (13):
- United States (13):
  - 1222.25.25009 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1222.25.25002 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1222.25.25003 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1222.25.25007 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 1222.25.25010 Boehringer Ingelheim Investigational Site, Austell, Georgia
  - 1222.25.25008 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1222.25.25012 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1222.25.25004 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1222.25.25011 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1222.25.25014 Boehringer Ingelheim Investigational Site, Seneca, South Carolina
  - 1222.25.25006 Boehringer Ingelheim Investigational Site, Knoxville, Tennessee
  - 1222.25.25005 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1222.25.25013 Boehringer Ingelheim Investigational Site, Richmond, Virginia

REFERENCES:
- [Derived] Feldman GJ, Bernstein JA, Hamilton A, Nivens MC, Korducki L, LaForce C. The 24-h FEV1 time profile of olodaterol once daily via Respimat(R) and formoterol twice daily via Aerolizer(R) in patients with GOLD 2-4 COPD: results from two 6-week crossover studies. Springerplus. 2014 Aug 9;3:419. doi: 10.1186/2193-1801-3-419. eCollection 2014. PMID 25187881

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, double-blind, double dummy, placebo- and active-controlled, 4 way crossover trial. The duration of each treatment period was 6 weeks with a 14 day washout period between treatments.
Groups:
- Placebo / Olo 5mcg / Olo 10mcg / Foradil 12mcg: Patients were administered placebo in the first period, Olodaterol 5 mcg qd in the second period, Olodaterol 10 mcg qd in the third period and Foradil 12 mcg bid in the fourth period. Olodaterol was administered via the Respimat inhaler, Foradil was administered via the Aerolizer inhaler.
- Olo 5mcg / Foradil 12mcg / Placebo / Olo 10mcg: Patients were administered Olodaterol 5mcg qd in the first period, Foradil 12 mcg bid in the second period, placebo in the third period and Olodaterol 10 mcg qd in the fourth period. Olodaterol was administered via the Respimat inhaler, Foradil was administered via the Aerolizer inhaler.
- Olo 10mcg / Placebo / Foradil 12mcg / Olo 5mcg: Patients were administered Olodaterol 10 mcg qd in the first period, placebo in the second period, Foradil 12 mcg bid in the third period and Olodaterol 5 mcg qd in the fourth period. Olodaterol was administered via the Respimat inhaler, Foradil was administered via the Aerolizer inhaler.
- Foradil 12mcg / Olo 10mcg / Olo 5mcg / Placebo: Patients were administered Foradil 12 mcg bid in the first period, Olodaterol 10 mcg qd in the second period, Olodaterol 5 mcg qd in the third period and placebo in the fourth period. Olodaterol was administered via the Respimat inhaler, Foradil was administered via the Aerolizer inhaler.
Period: Overall Study
Arm/Group | Placebo / Olo 5mcg / Olo 10mcg / Foradil 12mcg | Olo 5mcg / Foradil 12mcg / Placebo / Olo 10mcg | Olo 10mcg / Placebo / Foradil 12mcg / Olo 5mcg | Foradil 12mcg / Olo 10mcg / Olo 5mcg / Placebo
Started | 25 | 25 | 25 | 25
Completed | 20 | 22 | 21 | 24
Not Completed | 5 | 3 | 4 | 1
Not completed — Adverse Event | 2 | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Treated set, i.e. all treated patients.
Groups:
- Study Total: Total number of patients treated in the study. This was a randomised, double-blind, double dummy, placebo- and active-controlled, 4 way crossover trial. 99 patients were assigned randomly to one of 4 treatment sequences in which they received each of 4 treatments, two doses (5 microgram (mcg) or 10 mcg) of Olodaterol (Olo) once daily (qd) delivered via the Respimat inhaler or Foradil (Form) 12 mcg twice daily (bid) delivered via the Aerolizer inhaler or equivalent placebo delivered by Respimat Inhaler or Aerolizer Inhaler. The duration of each treatment period was 6 weeks with a 14 day washout period between treatments.
Arm/Group | Study Total
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: FEV1 Area Under Curve 0-12 h (AUC 0-12h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed in the morning of the first treatment visit, just prior to administration of the morning dose of randomized treatment. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FEV1 AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to am dose on the first day of treatment (baseline) and -30 min (zero time), 30 min, 60 min, 2 hour (h) , 3 h, 4 h, 6 h, 8 h, 10 h, 11 h 50 min relative to am dose after six weeks of treatment
Population: Full analysis set (FAS). FAS is defined as all patients with the baseline (pre-dose) date and any evaluable post-dosing data for the first co-primary endpoint FEV1AUC 0-12h.
Measure: Least Squares Mean (Standard Error); unit: Liter
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler or Aerolizer Inhaler.
- Olo 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Form 12 mcg Bid: Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler.
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 91 | 92 | 90 | 90
Liter | -0.022 (0.024) | 0.150 (0.024) | 0.152 (0.024) | 0.136 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a mixed model with center, treatment and period as fixed effects and patients within center as random effect; Mean Difference (Final Values) = 0.172, 95% CI [0.139 to 0.205], Standard Error of Mean 0.017 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.174, 95% CI [0.140 to 0.208], Standard Error of Mean 0.017 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.158, 95% CI [0.124 to 0.191], Standard Error of Mean 0.017 — Form 12 mcg bid minus Placebo

2. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-24 h (AUC 0-24h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random.FEV1 AUC 0-24h was calculated from 0-24 hours post-dose using the trapezoidal rule, divided by the observation time (24h) to report in litres.
Time Frame: 1 h and 10 min prior to am dose on the first day of the treatment (baseline) and -30 min, 30 min, 60 min, 2h, 3h, 4h, 6h, 8h, 10h, 11 hr 50 min,12 h 30 min, 13 h, 14 h, 22 h, 23 h, and 23 h 50 min relative to am dose after six weeks of treatment.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Groups:
- Placebo: Matching Placebo delivered by the Respimat resp. Aerolizer Inhaler.
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 91 | 92 | 90 | 90
Liter | -0.035 (0.024) | 0.110 (0.024) | 0.112 (0.024) | 0.121 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.145, 95% CI [0.114 to 0.176], Standard Error of Mean 0.016 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.147, 95% CI [0.116 to 0.179], Standard Error of Mean 0.016 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.156, 95% CI [0.125 to 0.187], Standard Error of Mean 0.016 — Form 12 mcg bid minus Placebo

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FEV1 AUC 0-3h was calculated from 0-3hours post-dose using the trapezoidal rule, divided by the observation time (3 h) to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and -30 min, 30 min, 60 min, 2 h , 3 h, relative to am dose after six weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 91 | 92 | 90 | 90
Liter | 0.004 (0.024) | 0.190 (0.025) | 0.202 (0.025) | 0.217 (0.025)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.186, 95% CI [0.149 to 0.223], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.198, 95% CI [0.162 to 0.235], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.213, 95% CI [0.176 to 0.250], Standard Error of Mean 0.019 — Form 12 mcg bid minus Placebo

4. Secondary Outcome: Peak FEV1 (0-3h) Response
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Peak values were obtained within 0 - 3 hours after the last am dose after six weeks of treatment. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 91 | 92 | 90 | 90
Liter | 0.076 (0.026) | 0.268 (0.026) | 0.273 (0.026) | 0.293 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.192, 95% CI [0.154 to 0.230], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.197, 95% CI [0.158 to 0.235], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.217, 95% CI [0.178 to 0.255], Standard Error of Mean 0.020 — Form 12 mcg bid minus Placebo

5. Secondary Outcome: Trough FEV1 Response
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Trough values were obtained 30 minutes prior to the last am dose of study drug after six weeks of treatment . Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 91 | 92 | 90 | 90
Liter | 0.012 (0.030) | 0.109 (0.030) | 0.115 (0.030) | 0.093 (0.030)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.097, 95% CI [0.045 to 0.148], Standard Error of Mean 0.026 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.103, 95% CI [0.051 to 0.155], Standard Error of Mean 0.026 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.080, 95% CI [0.028 to 0.132], Standard Error of Mean 0.026 — Form 12 mcg bid minus Placebo

6. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-12 Hours (AUC 0-12h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FVC AUC 0-12h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: as for outcome 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 91 | 92 | 90 | 90
Liter | -0.032 (0.040) | 0.219 (0.040) | 0.214 (0.040) | 0.203 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.251, 95% CI [0.195 to 0.306], Standard Error of Mean 0.028 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.246, 95% CI [0.190 to 0.302], Standard Error of Mean 0.028 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.235, 95% CI [0.179 to 0.291], Standard Error of Mean 0.028 — Form 12 mcg bid minus Placebo

7. Secondary Outcome: FVC Area Under Curve 12-24 Hours (AUC 12-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FVC AUC 12-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 h and 10 min prior to am dose on the first day of treatment (baseline) and 12 h 30 min, 13 h, 14 h, 22 h, 23 h, and 23 h 50 min relative to am dose after six weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 91 | 92 | 90 | 90
Liter | -0.078 (0.041) | 0.083 (0.041) | 0.079 (0.041) | 0.144 (0.041)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.161, 95% CI [0.101 to 0.222], Standard Error of Mean 0.031 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.157, 95% CI [0.096 to 0.218], Standard Error of Mean 0.031 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.223, 95% CI [0.162 to 0.284], Standard Error of Mean 0.031 — Form 12 mcg bid minus Placebo

8. Secondary Outcome: FVC Area Under Curve 0-24 Hours (AUC 0-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FVC AUC 0-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 h and 10 min prior to am dose on the first day of treatment (baseline) and -30 min, 30 min, 60 min, 2h, 3h, 4h, 6h, 8h, 10h, 11 hr 50 min,12 h 30 min, 13 h, 14 h, 22 h, 23 h, and 23 h 50 min relative to am dose after six weeks of treatment.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 91 | 92 | 90 | 90
Liter | -0.055 (0.039) | 0.151 (0.039) | 0.147 (0.039) | 0.174 (0.039)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.206, 95% CI [0.155 to 0.258], Standard Error of Mean 0.026 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.202, 95% CI [0.150 to 0.255], Standard Error of Mean 0.027 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.229, 95% CI [0.176 to 0.281], Standard Error of Mean 0.027 — Form 12 mcg bid minus Placebo

9. Secondary Outcome: Peak FVC (0-3h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Peak FVC was obtained within 0 - 3 hours after the last am dose of study drug after 6 weeks of treatment. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 91 | 92 | 90 | 90
Liter | 0.138 (0.043) | 0.436 (0.043) | 0.440 (0.043) | 0.475 (0.043)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.299, 95% CI [0.233 to 0.365], Standard Error of Mean 0.034 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.302, 95% CI [0.236 to 0.369], Standard Error of Mean 0.034 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.338, 95% CI [0.271 to 0.405], Standard Error of Mean 0.034 — Form 12 mcg bid minus Placebo

10. Secondary Outcome: Trough FVC Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Trough values were obtained 30 minutes prior to the last am dose of study drug after six weeks of treatment . Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 91 | 92 | 90 | 90
Liter | -0.007 (0.053) | 0.125 (0.053) | 0.133 (0.054) | 0.141 (0.054)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0163, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.132, 95% CI [0.024 to 0.239], Standard Error of Mean 0.055 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0118, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.139, 95% CI [0.031 to 0.247], Standard Error of Mean 0.055 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p = 0.0076, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.148, 95% CI [0.040 to 0.256], Standard Error of Mean 0.055 — Form 12 mcg bid minus Placebo

11. Primary Outcome: FEV1 Area Under Curve 12-24h (AUC 12-24h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed in the morning of the first treatment visit, just prior to administration of the morning dose of randomized treatment. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FEV1 AUC 12-24h was calculated from 12-24 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: as for outcome 7
Population: Full analysis set (FAS).
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 91 | 92 | 90 | 90
Liter | -0.048 (0.025) | 0.069 (0.025) | 0.072 (0.025) | 0.107 (0.025)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.118, 95% CI [0.082 to 0.154], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.120, 95% CI [0.084 to 0.157], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.155, 95% CI [0.119 to 0.191], Standard Error of Mean 0.018 — Form 12 mcg bid minus Placebo

12. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG
Description: Clinical relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG. New abnormal findings or worsenings of baseline conditions were reported as Adverse Events related to treatment (cardiac disorders and investigations).
Time Frame: 6 weeks
Measure: Number; unit: participants
Groups:
- Olo 5 mcg: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Form 12 mcg: Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler.
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg | Form 12 mcg
Number analyzed (Participants) | 94 | 93 | 95 | 93
participants
  Bundle branch block right | 0 | 0 | 1 | 0
  ECG QT prolonged | 0 | 0 | 1 | 0
  Tachycardia | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg | Form 12 mcg
Serious Adverse Events (participants affected / at risk) | 3/94 | 4/93 | 3/95 | 5/93
Other Adverse Events (participants affected / at risk) | 9/94 | 9/93 | 12/95 | 7/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | Olo 5 mcg (N=93) | Olo 10 mcg (N=95) | Form 12 mcg (N=93)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | Olo 5 mcg (N=93) | Olo 10 mcg (N=95) | Form 12 mcg (N=93)
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 5 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 7 | 2

LIMITATIONS AND CAVEATS:
1. Safety assessments are potentially confounded by both crossover and long washout periods
2. Comparisons of active groups for the 12 to 24 hr period overestimate the effect of Foradil (sleeping period causing an overestimation of AUC)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication